CLINICAL TRIAL: NCT00212225
Title: Risk Factors for Gastric Disease in Pediatric H. Pylori
Brief Title: Risk Factors for Gastric Disease in Pediatric Helicobacter Pylori (H. Pylori)
Status: Completed | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Other Study IDs: DK53708 (completed)
Record Dates: First submitted 2005-09-20; First posted 2005-09-21 (Estimated); Last update posted 2010-01-13 (Estimated); Status verified 2010-01

CONDITIONS: Helicobacter Infections; Gastritis; Peptic Ulcer
Keywords: gastric disease; H. pylori; children; Helicobacter pylori; child; epidemiology
MeSH Terms: conditions — Helicobacter Infections; Gastritis; Peptic Ulcer; Stomach Diseases

SUMMARY:
Helicobacter pylori (Hp) is a major cause of chronic-active gastritis and primary duodenal ulcers, and is strongly linked to gastric cancer. Most Hp infections worldwide are acquired in childhood. Why some individuals develop symptomatic disease is unclear and, until recently, no studies critically evaluated the role of pediatric Hp strains and/or host factors in disease outcomes. Over the past 5 years of National Institutes of Health (NIH) funding, 486 children from Atlanta, Cleveland, and Miami were enrolled; 184 (38%) were Hp-infected. Race (African American) and younger age, in conjunction with Hp strains expressing cagA and vacAs1B, were shown to be risk factors for both esophageal and gastric disease, suggesting a different disease paradigm from Hp-infected adults. Using the updated Sydney system, the investigators demonstrated a histopathologic spectrum in children, which included novel observations of atrophic gastritis with intestinal metaplasia.

Overall hypothesis for competitive renewal: disease manifestations in Hp-infected children are influenced by specific host factors (i.e., race, immune phenotype), environmental exposures, and specific virulence factors of infecting Hp strains.

Specific aims:

1. Using well defined cases and controls, further characterize specific host factors and environmental exposures contributing to symptomatic childhood infection emphasizing targeted enrollment in specific age, gender and demographic strata to facilitate detection of significant differences not attained previously and follow-up of 2 established specific cohorts to ascertain immune response natural history.
2. Utilize gene-array technology for the whole Hp genome assessment and bacterial gene expression of specific virulence determinants associated with pediatric Hp strains.
3. Further characterize the host immunologic and mucosal response in Hp-infected children.

Hp-infected symptomatic endoscopy cases at the investigators' established 3 clinical centers of high, moderate and low Hp prevalence will be compared with age-matched Hp-infected asymptomatic and uninfected symptomatic controls. Two geographically and demographically distinct centers have been added to provide additional geographic and subject representativeness to the patient cohort. The updated Sydney system will be employed to assess gastric histopathology severity and phenotype in newly enrolled cases in specific age, gender and demographic strata and follow-up of the two "novel" cohorts established in the past 5 years: a) atrophic gastritis; and b) esophageal and gastric disease groups enabling a comprehensive, multivariate evaluation of the natural history of Hp-infected children in two distinct disease paradigms.

Using molecular methods (multiplex [MP]-PCR, RT-PCR) and a micro ELISPOT assay on peripheral blood mononuclear cells (PBMCS), Th1, Th2, Th3 or balanced Th1/Th2 response will be determined to further characterize the Hp-infected child's immune response phenotype. The investigators propose to further their previous work with critically lacking studies from a multivariate approach, leading to a better understanding of the gastroduodenal disease sequelae and overall pathobiology of Hp infection in humans.

DETAILED DESCRIPTION:
Discovered in 1982 as a cause of gastroduodenal ulceration, Helicobacter pylori (Hp) is the major cause of gastritides (e.g. chronic-active) and primary duodenal ulcers in adults and children. [Warren, 1983 #1180; Whitney, 2000 #1345; Ashorn, 1995 #1179; Asante, 1997 #1173; Drumm, 1987 #355; Czinn, 1986 #101; Drumm, 1988 #1096; Ernst, 2000 #1351; Goggin, 1998 #986; Torres, 2000 #1346] Infection with Hp, particularly in susceptible persons, is also strongly linked to gastric adenocarcinoma cancer and mucosal-associated lymphoid tissue-type (MALT) lymphomas. [Uemura, 2001 #1409; Alexander, 2000 #1232; Alm, 1999 #1038; Blaser, 1995 #757; Correa, 1990 #1523; El-Omar, 2000 #1272] The majority of infections worldwide are acquired in childhood. In the United States, minority populations (African Americans, Hispanics) have increased seroprevalence rates in all age groups. [Fontham, 1995 #139; Gold, 2001 #1422; Graham, 1991 #235; Staat, 1996 #190; Smoak, 1994 #618] Consensus guidelines for pediatric Hp infection were first published in 1999, yet there remains an overwhelming paucity of information regarding both the epidemiology of pediatric Hp infection and associated diseases. [Gold, 2000 #1347; Drumm, 2000 #1123; Sherman, 1999 #1129; Hunt, 1998 #353] It is not known why some Hp-infected children develop symptoms, and mechanisms accounting for differences in the inflammatory response and disease in Hp-infected children are uncharacterized. Using a multicenter study approach to test our hypothesis, this proposal will provide an in depth examination of the association between host factors, Hp strain genotype, and the severity of gastric inflammatory response in children. Variation between age, race/ethnicity, medical/environmental exposures, socioeconomic status and geographic regions and their effects on disease phenotype in children will be investigated. These studies will address unanswered questions about the earliest stages in the pathobiology of Hp infection that are essential to improve our ability to manage this infection in children, and potentially, identify and understand "at risk groups" to prevent more severe disease sequelae in adults. Understanding the evolution of the host response to Hp infection is needed to develop prevention strategies or new therapies, and allow a better definition of the pathobiology of this human pathogen that causes significant morbidity, suffering, and economic impact in our society.

In our 5 years of NIH funding, we enrolled a cohort of 486 children from 3 sites (Atlanta, Cleveland, Miami); 184 (38%) were Hp-infected. We made novel observations regarding environmental exposures, pilot validation of a symptom assessment instrument, pediatric Hp strain genotype/disease phenotype relationships, and disease paradigms not previously described in the pediatric population; i.e., atrophic gastritis and intestinal metaplasia associated with Hp infection. Overall hypothesis for competitive renewal: gastroduodenal disease (e.g., duodenal ulcer) in Hp-infected children is associated with specific host factors (i.e., race/ethnicity), environmental exposures, and infection by Hp strains carrying specific virulence genes contained within the cag pathogenicity island. These combined factors drive either a predominant Th2 gastric mucosal response with antral predominant severe mucosal inflammation (i.e., ulcer disease) or a Th1 response resulting in a more chronic, corpus-predominant inflammatory infiltrate (i.e., atrophy).

Specific aims:

Aim 1: Further characterize specific host factors and environmental exposures contributing to symptomatic childhood infection by emphasizing targeted enrollment of patients from multiple centers in specific age, gender and demographic strata to facilitate detection of significant differences in symptomatic and asymptomatic Hp-infected children not attained previously and follow-up of 2 established specific cohorts to ascertain immune response natural history.

Aim 2: Utilize gene-array technology for whole genome assessment of bacterial virulence genes and specific bacterial gene expression to allow characterization of virulence proteins associated with pediatric Hp infection. The Hp isolated from the prospectively enrolled infected children (cases) in Aim 1, Hp strains obtained in follow-up of the two established cohorts who remain infected, as well as a retrospective analysis of 125 banked pediatric isolates linked to clinical, demographic and epidemiological data will be characterized. Specific emphasis will be on the analysis of isolates found in the following three disease categories: ulcers, gastritis, atrophic gastritis.

Aim 3: Further characterize the gastric mucosal host inflammatory response in Hp-infected children.

The Updated Sydney system will be applied to assess severity of gastric histopathology, and immunohistochemistry performed on formalin-fixed, paraffin embedded tissues to phenotype mucosal disease (i.e., character, severity) in newly enrolled cases in specific age, gender and demographic strata and the two "novel" cohorts established in our previous studies; i) atrophic gastritis cohort; ii) esophageal and gastric disease cohort, affording insight into the natural history of the immune response in Hp-infected children in two different disease paradigms. Both molecular methods and a novel micro ELISPOT performed on PBMCS and gastric T-cells to determine Th1, Th2 or balanced Th1/Th2 response will be used to further characterize the Hp-infected child's immune phenotype. During the latter 2 years of the proposed studies, PBMC chemokine response will then be compared to the mucosal/cellular response using RT-PCR and gene array. The data obtained from aims 1 and 3 will be integrated with that obtained in aim 2 (Hp-strain genotype) in order to develop a model to predict disease outcome based on host demographics, strain type and inflammatory/immune response. These studies are critical to understand and better predict the gastroduodenal disease sequelae and overall pathobiology of Hp infection in humans.

ELIGIBILITY:
Inclusion Criteria:

* Using the power determinations for age, gender and demographic characteristics, the investigators will screen all patients undergoing diagnostic upper endoscopy at:

  * Children's Healthcare of Atlanta (Egleston and Scottish Rite Children's Hospitals), Atlanta, GA
  * Rainbow Babies and Children's Hospital, Cleveland, OH
  * Miami Children's Hospital, Miami, FL.
* Patients will be enrolled over the first 3 years of the study, and then based on interim univariate analysis. The investigators also will perform follow-up evaluations (i.e., clinically-indicated) on the two novel cohorts identified during the first 5 years of funding:

  * the atrophic gastritis Hp-infected cohort
  * the esophagitis/gastritis cohort, in order to assess the natural history of gastroduodenal inflammation in the Hp-infected child.

Exclusion Criteria:

* Patients who have taken antibiotics within one month of endoscopy will be excluded, as preceding antibiotic therapy will confound ability to determine Hp infection status.
* In the previous five years, the investigators initially eliminated children taking proton pump inhibitors (PPIs) (e.g., omeprazole); Na+/H+ ATPase channel inhibitors. PPIs have a minimum inhibitory concentration (MIC) against Hp in vitro, and therefore may reduce the overall bacterial load, diminishing the ability to detect infection, and resolve gastroduodenal mucosal inflammation, confounding characterization of cellular host response to Hp infection. However, due to the pervasive use of PPIs in the pediatric population, and the exclusion of potential cases, the investigators improved their culture sensitivity techniques and are able to successfully detect the organism in the setting of a child on a PPI. This will be taken into account when characterizing the gastric mucosal inflammatory phenotype and comparative analyses are performed.

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 755 (Estimated)
Dates: Start 1997-10; Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin D. Gold, M.D., Principal Investigator — Emory University
Locations (3):
- United States (3):
  - Miami Children's Hospital; Division of Pediatric Gastroenterology, Miami, Florida
  - Emory University School of Medicine; Emory Children's Center, Atlanta, Georgia
  - Case Western Reserve University; Rainbow Babies and Children's Hospital, Cleveland, Ohio